CLINICAL TRIAL: NCT04351893
Title: Craniofacial Microsomia: Accelerating Understanding of the Significance and Etiology
Acronym: CAUSE
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Children's Hospital Los Angeles (Other); Children's Hospital of Philadelphia (Other); University of North Carolina, Chapel Hill (Other); Pontificia Universidad Javeriana (Other); Universidad Icesi (Other); Hospital Nacional Edgardo Rebagliati Martins (Other); Instituto de Investigación Hospital Universitario La Paz (Other); Clinica Comfamiliar Risaralda (Unknown)
Responsible Party: Principal Investigator, Carrie Heike, Professor, Seattle Children's Hospital
Other Study IDs: 17-601-E
Record Dates: First submitted 2020-04-11; First posted 2020-04-17 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Microtia; Microtia-Anotia; Craniofacial Microsomia; Goldenhar Syndrome; OAVS; OAV Syndrome; Hemifacial Microsomia
MeSH Terms: conditions — Congenital Microtia; Microtia-Anotia; Goldenhar Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants are asked for blood or saliva. If a participant is having a surgery, tissue that would otherwise be discarded would also be requested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CAUSE study is a multicenter study, with domestic (n=4) and international (n=6) study sites. Children and young adults (ages 0-18) who have microtia and/or craniofacial microsomia and their parents are invited to participate. Children and parents are asked to provide a DNA sample (blood or saliva) and are asked to upload a few photos of their face. Parents are asked a short interview. Participants are able to participate from home or at one of four domestic sites.

ELIGIBILITY:
INCLUSION:

Cases:

* Participant with CFM is 0-18 years of age
* Participant has diagnosis of at least one of the following conditions:

  * Microtia
  * Anotia
  * Facial asymmetry AND preauricular tag(s)
  * Facial asymmetry AND facial tag(s)
  * Facial asymmetry AND epibulbar dermoid
  * Facial asymmetry AND macrostomia (i.e., lateral cleft)
  * Preauricular tag AND epibulbar dermoid
  * Preauricular tag AND macrostomia
  * Facial Tag AND epibulbar dermoid
  * Macrostomia AND epibulbar dermoid
* Participant's parent or legal guardian has provided written informed consent prior to enrollment into study (for participants younger than 18 years of age).
* Participant speaks a language in which they are eligible for consent at their enrolling site

Parents:

* Parent participant is the biological parent of a case participant already eligible and participating in the CAUSE study. Non-genetic parents will be interviewed about their child's known prenatal and genetic family history but will not be asked to provide DNA or have facial photographs taken.
* Participant speaks a language in which they are eligible for consent at their enrolling site

Other relatives:

* Other relatives participants, of any age, are related biologically to a case participant already eligible and participating in the CAUSE study from a multiplex family (multiple affected individuals with CFM).
* Participant speaks a language in which they are eligible for consent at their enrolling site

EXCLUSION:

Cases:

* Participant is diagnosed with a known syndrome that involves microtia and underdevelopment of the jaw (Townes-Brocks, Treacher-Collins, Branchiootorenal, Nager, or Miller syndromes).
* Participant has abnormal chromosome studies (karyotype).
* Participant has mandibular asymmetry due to deformational plagiocephaly or torticollis.

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All CFM cases, their parents, and their relatives regardless of their sex, race, or ethnicity. The prospective case samples will likely be drawn from outpatient clinics and medical centers, as well as CFM-related social medial networks.
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Identify Genetic Variants | Through study completion, an average of 1 year.
  To identify genetic variants related to the CFM spectrum using whole genome sequencing

SECONDARY OUTCOMES:
Characterize phenotype | Through study completion, an average of 1 year.
  To characterize the detailed phenotype in individuals with CFM
Characterize markers | Through study completion, an average of 1 year.
  To characterize ancestry markers in individuals with CFM
Coding and non-coding variants | Through study completion, an average of 1 year.
  To assess coding and non-coding variants in selected candidate genes in individuals with CFM

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Heike, MD, MS, Principal Investigator — Seattle Children's Hospital
Locations (10):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- Colombia (4):
  - Pontificia Universidad Javeriana, Bogotá
  - ICESI, Cali
  - Pontificia Universidad Javeriana, Cali
  - Clínica Comfamiliar Risaralda, Pereira
- Hospital Edgardo Rebagliati Martins, Lima, Peru
- Instituto de Genética Médica y Molecular (INGEMM), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share, as CFM is a rare disease and could be potentially identifiable.